CLINICAL TRIAL: NCT05949541
Title: Study of Efficacy of Everolimus Combined With First-line Endocrine Therapy for HR+/HER2- (Open, Randomized, Phase II )
Brief Title: Efficacy of Everolimus Combined With First-line Endocrine Therapy for HR+/HER2- SNF1-subtype Advanced Breast Cancer
Acronym: BCTOP-L-M01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N062
Record Dates: First submitted 2023-07-09; First posted 2023-07-18 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Advanced Breast Cancer
Keywords: luminal breast cancer; advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; dalpiciclib; Aromatase Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm-A (Experimental): Everolimus + CDK4/6 inhibitor+ Endocrine therapy group:
  Everolimus, 10mg po. qd; Dalpiciclib 125mg po. qd. for 3 weeks, followed by 1 week off, 4 weeks as a cycle.
  Aromatase inhibitors (Letrozole/Anastrozole/Exemestane), po. qd. at specific doses (Letrozole 2.5mg/day; Anastrozole 1mg/day, Exemestane 25mg/day); Or Fluvestrant, 500mg im. q28d, (Extra 500mg given after 2 weeks of first dose); Premenopause participants: Goserelin 3.6mg, subcutaneously, once every 4 weeks.
  Interventions: Drug: Everolimus 10 mg; Drug: CDK4/6 Inhibitor SHR6390; Drug: Aromatase inhibitor and Fulvestrant combined with CDK4/6 inhibitors
- Arm-B (Active Comparator): CDK4/6 inhibitor+ Endocrine therapy group:
  Dalpiciclib 125mg po. qd. for 3 weeks, followed by 1 week off, 4 weeks as a cycle.
  Aromatase inhibitors (Letrozole/Anastrozole/Exemestane), po. qd. at specific doses (Letrozole 2.5mg/day; Anastrozole 1mg/day, Exemestane 25mg/day); Or Fluvestrant, 500mg im. q28d, (Extra 500mg given after 2 weeks of first dose); Premenopause participants: Goserelin 3.6mg, subcutaneously, once every 4 weeks.
  Interventions: Drug: CDK4/6 Inhibitor SHR6390; Drug: Aromatase inhibitor and Fulvestrant combined with CDK4/6 inhibitors

INTERVENTIONS:
Drug: Everolimus 10 mg — Everolimus is a kind of mTOR inhibitor which has been approved to use in several kinds of cancers, especially in metastatic breast cancer.
  Other Names: Afinitor
  Arms: Arm-A
Drug: CDK4/6 Inhibitor SHR6390 — Dalpiciclib (SHR6390) is a kind of CDK4/6 inhibitor that has demonstrated tolerability and preliminary clinical activity in patients with heavily pretreated hormone receptor-positive, HER2-negative advanced breast cancer.
  Other Names: Dalpiciclib
Drug: Aromatase inhibitor and Fulvestrant combined with CDK4/6 inhibitors — Endocrine therapy combined with CDK4/6 inhibitors is the standard first-line therapy for advanced luminal breast cancer. Investigators choose endocrine therapy including Letrozole, Anastrozole, Exemestane, and Fulvestrant. Postmenopausal participants should use Goserelin.
  Other Names: Endocrine therapy

SUMMARY:
This is a randomized, controlled, open-label, phase II study to explore the efficacy and safety of Everolimus in combination with standard first-line endocrine therapy for the HR+/ HER2-SNF1 subtype of advanced breast cancer. The study was used to explore the efficacy of Everolimus in combination with standard endocrine therapy.

DETAILED DESCRIPTION:
A total of 584 patients with luminal breast cancer who received surgery in the breast surgery Department of the Affiliated Cancer Hospital of Fudan University were collected in the early stage. All patients could be divided into four categories, namely SNF1 (classical luminal type), SNF2 (immune-mediated type), SNF1 (proliferative type), and SNF4 (receptor tyrosine kinase-driven type), through clustering by the SNF algorithm. SNF1 (classical luminal type): The transcriptional component type is dominated by PAM50 LumA, with high PIK3CA mutation and low TP53 mutation. By combining artificial intelligence based on H&E pathological sections with deep learning methodology, molecular typing can be effectively distinguished. Prior to enrollment, the patient's primary lesion or metastasis was classified by molecular classification based on the H&E section combined with digital pathology, and SNF1 was confirmed to be considered for subsequent enrollment.

Receivers will be randomly assigned 1:1 to either Everolimus plus Standard Endocrine therapy (study group) or Standard Endocrine therapy (control group).

Treatment will continue until disease progression, intolerable toxicity, informed withdrawal, or death from any cause.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to meet all of the following conditions

  * Patients must be ≥18 and ≤ 75 years of age;
  * Pathologically confirmed breast cancer is HR+/HER2- breast cancer (IHC ER >10%, or/and PR>10%, HER 0 OR +, if HER2++, FISH negative);
  * SNF1 subtype definition: SNF1 subtype confirmed by digital pathology of H&E sections;
  * Locally advanced breast cancer (radical local therapy is not possible) or metastatic breast cancer (without using adjuvant CDK4/6 inhibitors in the past, or one year after adjuvant CDK4/6 inhibitor therapy has ended);
  * No prior therapy (chemotherapy, targeted therapy, etc.) for advanced or metastatic breast cancer;
  * Patients with at least one measurable lesion that has not previously received radiation therapy and can be evaluated repeatedly according to RECIST 1.1;
  * The functions of the main organs are basically normal, and the following conditions are met:

    1. Blood routine examination standards should meet: HB≥90g/L (no blood transfusion within 14 days); ANC≥1.5×109/L; PLT≥75×109/L;
    2. Biochemical examination shall meet the following standards: TBIL≤1.5×ULN (upper limit of normal value); ALT and AST≤3 x ULN; In case of liver metastasis, ALT and AST≤5×ULN; Serum Cr ≤1.5×ULN, endogenous creatinine clearance > 50ml/min (Cockcroft-Gault formula);
  * ECOG performance status 0 or 1; The expected survival is more than 3 months;
  * Fertile female is required to use a medically approved contraceptive during study treatment and for at least 3 months after the last use of the study drug;
  * Patients voluntarily join the study, sign the informed consent, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Patients with any of the following conditions were excluded from the study

  * Patients with central nervous system metastasis out of control (symptoms need to use glucocorticoids or mannitol).
  * A history of clinically significant or uncontrolled heart disease, including congestive heart failure, angina pectoris, myocardial infarction within the last 6 months, or ventricular arrhythmia;
  * Radiotherapy, chemotherapy, surgery, other targeted therapy and immunotherapy for advanced HR+/HER2- breast cancer within 4 weeks prior to first administration of drugs used in this study.
  * Pregnant or lactating patients;
  * Other malignancies within the previous 3 years, excluding cured skin basal cell carcinoma and cervical carcinoma in situ;
  * Significant comorbid medical conditions, including mental illnesses that the investigator or sponsor believes would adversely affect the patient's participation in the study;
  * Allergic physique, or known allergic history of the drug components of this program; Or allergic to other monoclonal antibodies;
  * The investigator does not consider the patient suitable for participation in any other circumstances of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Approximately 5 years
  The interval from randomization until the first occurrence of disease progression (according to RECIST 1.1) or death from any cause, which ever occurs first.

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | Approximately 5 years
  CBR is the total percentage of participants who achieved a complete response, partial response, or had stable disease for 6 months or more.
Objective Response Rate (ORR) | Approximately 5 years
  ORR is defined as the proportion of participants who have a complete response (CR) or partial response (PR) based on BICR and investigator assessment using RECIST 1.1.
Overall Survival (OS) | Approximately 5 years
  OS is defined as the time from randomisation until the date of death due to any cause.
Safety and tolerability | Approximately 5 years
  Number of adverse events according to NCI-CTCAE Version 5.0 per each treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, MD,PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China